CLINICAL TRIAL: NCT02334787
Title: A Single-center, Placebo-controlled, Randomized, Double-blind, Parallel-group Comparison Trial to Assess the Safety and Pharmacokinetics of OPA-15406 Ointment in Healthy Adult Male Subjects (Phase 1 Trial)
Brief Title: A Phase 1 Trial of OPA-15406 Ointment in Healthy Adult Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 271-14-001
Record Dates: First submitted 2015-01-05; First posted 2015-01-08 (Estimated); Results first posted 2016-10-03 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2016-08

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- 0.3% OPA-15406 in a single administration period (Experimental): 32 subjects were randomly allocated to 4 treatment groups (8 subjects per dose). In a single administration period, subjects were treated with assigned0.3% OPA-15406 ointment assessed until 48 hours postdose.
  Interventions: Drug: 0.3% OPA-15406 Ointment
- 1% OPA-15406 in a single administration period (Experimental): 32 subjects were randomly allocated to 4 treatment groups (8 subjects per dose). In a single administration period, subjects were treated with assigned 1% OPA-15406 ointment assessed until 48 hours postdose.
  Interventions: Drug: 1% OPA-15406 Ointment
- 3% OPA-15406 in a single administration period (Experimental): 32 subjects were randomly allocated to 4 treatment groups (8 subjects per dose). In a single administration period, subjects were treated with assigned 3% OPA-15406 ointment assessed until 48 hours postdose.
  Interventions: Drug: 3% OPA-15406 Ointment
- Placebo in a single administration period (Placebo Comparator): 32 subjects were randomly allocated to 4 treatment groups (8 subjects per dose). In a single administration period, subjects were treated with assigned placebo ointment assessed until 48 hours postdose.
  Interventions: Drug: Placebo Ointment
- 0.3% OPA-15406 in the multiple administration period (Experimental): In the multiple administration period, same subjects were treated with assigned 0.3% OPA-15406 ointment twice daily for 14 days and assessed until 48 hours post dose.
  Interventions: Drug: 0.3% OPA-15406 Ointment
- 1% OPA-15406 in the multiple administration period (Experimental): In the multiple administration period, same subjects were treated with assigned 1% OPA-15406 ointment twice daily for 14 days and assessed until 48 hours post dose.
  Interventions: Drug: 1% OPA-15406 Ointment
- 3% OPA-15406 in the multiple administration period (Experimental): In the multiple administration period, same subjects were treated with assigned 3% OPA-15406 ointment twice daily for 14 days and assessed until 48 hours post dose.
  Interventions: Drug: 3% OPA-15406 Ointment
- Placebo in the multiple administration period (Experimental): In the multiple administration period, same subjects were treated with assigned OPA-15406 ointment placebo twice daily for 14 days and assessed until 48 hours post dose.
  Interventions: Drug: Placebo Ointment

INTERVENTIONS:
Drug: 0.3% OPA-15406 Ointment — 32 subjects were randomly allocated to 4 treatment groups (8 subjects per dose). In a single administration period, subjects were treated with assigned 0.3 % OPA-15406 ointment assessed until 48 hours postdose. In the multiple administration period, same subjects were treated with assigned 0.3% OPA-15406 ointment twice daily for 14 days and assessed until 48 hours post dose.
  Other Names: OPA-15406 Ointment
  Arms: 0.3% OPA-15406 in a single administration period; 0.3% OPA-15406 in the multiple administration period
Drug: 1% OPA-15406 Ointment — 32 subjects were randomly allocated to 4 treatment groups (8 subjects per dose). In a single administration period, subjects were treated with assigned 1 % OPA-15406 ointment assessed until 48 hours postdose. In the multiple administration period, same subjects were treated with assigned 1% OPA-15406 ointment twice daily for 14 days and assessed until 48 hours post dose
  Other Names: OPA-15406 Ointment
  Arms: 1% OPA-15406 in a single administration period; 1% OPA-15406 in the multiple administration period
Drug: 3% OPA-15406 Ointment — 32 subjects were randomly allocated to 4 treatment groups (8 subjects per dose). In a single administration period, subjects were treated with assigned 3 % OPA-15406 ointment assessed until 48 hours postdose. In the multiple administration period, same subjects were treated with assigned 3% OPA-15406 ointment twice daily for 14 days and assessed until 48 hours post dose.
  Other Names: OPA-15406 Ointment
  Arms: 3% OPA-15406 in a single administration period; 3% OPA-15406 in the multiple administration period
Drug: Placebo Ointment — 32 subjects were randomly allocated to 4 treatment groups (8 subjects per dose). In a single administration periodriod, subjects were treated with assigned placebo ointment assessed until 48 hours postdose. In the multiple administration period, same subjects were treated with assigned placebo ointment twice daily for 14 days and assessed until 48 hours post dose.
  Arms: Placebo in a single administration period; Placebo in the multiple administration period

SUMMARY:
To assess the safety (especially skin findings) and pharmacokinetics by applying 0.3%, 1%, or 3% formulation of 5g OPA-15406 ointment to a 1000 cm2 area as a single-dose and as a multiple-dose twice daily for 2 weeks in Japanese healthy adult male subjects.

ELIGIBILITY:
Inclusion Criteria:

* BMI = Body weight (kg) / [Height (m)]2: at least 18.5 and less than 25.0
* Judged by the investigator or subinvestigator to be healthy based on test results at screening and prior to administration on Day 1 of the treatment period

Exclusion Criteria:

* Findings (sunburn, abrasions, tattoos, etc) on the back that affect the evaluation of the safety of the skin
* Judged by the investigator or subinvestigator as inappropriate to participate in this trial for any other reasons

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2015-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hiroaki Ono, Mr, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (1):
- Kanto Region, Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- 0.3% OPA-15406 Ointment: In a single administration period and the multiple administration period, same subjects were treated with assigned 0.3% OPA-15406 ointment.
- 1% OPA-15406 Ointment: In a single administration period and the multiple administration period, same subjects were treated with assigned 1% OPA-15406 ointment.
- 3% OPA-15406 Ointment: In a single administration period and the multiple administration period, same subjects were treated with assigned 3% OPA-15406 ointment.
- Placebo: In a single administration period and the multiple administration period, same subjects were treated with assigned placebo ointment.
Period: Overall Study
Arm/Group | 0.3% OPA-15406 Ointment | 1% OPA-15406 Ointment | 3% OPA-15406 Ointment | Placebo
Started | 8 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.3% OPA-15406 Ointment | 1% OPA-15406 Ointment | 3% OPA-15406 Ointment | Placebo | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 8 | 8 | 32
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.9 (7.2) | 28.3 (7.6) | 30.5 (6.7) | 29.5 (6.3) | 30.0 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 8 | 8 | 8 | 8 | 32
Region of Enrollment [Number; unit: participants]
  Japan | 8 | 8 | 8 | 8 | 32

OUTCOME MEASURES:

1. Primary Outcome: Cmax of OPA-15406 in a Single Administration Period
Description: We measure the plasma concentration of OPA-15406 at Day 1 by applying 0.3%, 1%, or 3% formulation of OPA-15406 ointment as a single dose. We assess the Cmax of OPA-15406.
Time Frame: Baseline, 2 ,3, 4, 8, 10, 12, 16, 24 and 48 hr
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- 0.3% OPA-15406 Ointment in a Single Administration Period: 32 subjects were randomly allocated to 4 treatment groups (8 subjects per dose). In a single administration period, subjects were treated with assigned0.3％OPA-15406 ointment assessed until 48 hours postdose.
- 1% OPA-15406 Ointment in a Single Administration Period: 32 subjects were randomly allocated to 4 treatment groups (8 subjects per dose). In a single administration period, subjects were treated with assigned 1% OPA-15406 ointment assessed until 48 hours postdose.
- 3% OPA-15406 Ointment in a Single Administration Period: 32 subjects were randomly allocated to 4 treatment groups (8 subjects per dose). In a single administration period, subjects were treated with assigned 3% OPA-15406 ointment assessed until 48 hours postdose.
Arm/Group | 0.3% OPA-15406 Ointment in a Single Administration Period | 1% OPA-15406 Ointment in a Single Administration Period | 3% OPA-15406 Ointment in a Single Administration Period
Number analyzed (Participants) | 8 | 8 | 8
ng/mL | 0.508 (0.304) | 0.838 (0.531) | 1.61 (0.835)

2. Primary Outcome: Cmax of OPA-15406 in the Multiple Administration Period
Description: We measure the plasma concentration of OPA-15406 from Day 1 to Day 14 by applying 0.3%, 1%, or 3% formulation of OPA-15406 ointment as multiple doses twice daily for 2 weeks. We assess the AUC12h x of OPA-15406.
Time Frame: Baseline, 2 ,3, 4, 8, 10, 12, 16, 24 and 48 hrs at Day 14
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- 0.3 % OPA-15406 Ointment in the Multiple Administration Period: In the multiple administration period, same subjects were treated with assigned 0.3％OPA-15406 ointment twice daily for 14 days and assessed until 48 hours post dose.
- 1 % OPA-15406 Ointment in the Multiple Administration Period: In the multiple administration period, same subjects were treated with assigned 1％OPA-15406 ointment twice daily for 14 days and assessed until 48 hours post dose.
- 3% OPA-15406 Ointment in the Multiple Administration Period: In the multiple administration period, same subjects were treated with assigned 3％OPA-15406 ointment twice daily for 14 days and assessed until 48 hours post dose.
Arm/Group | 0.3 % OPA-15406 Ointment in the Multiple Administration Period | 1 % OPA-15406 Ointment in the Multiple Administration Period | 3% OPA-15406 Ointment in the Multiple Administration Period
Number analyzed (Participants) | 8 | 8 | 8
ng/mL | 0.506 (0.348) | 0.795 (0.208) | 1.65 (0.462)

3. Secondary Outcome: AUC12h of OPA-15406 in a Single Administration Period
Description: We measure the plasma concentration of OPA-15406 at Day 1 by applying 0.3%, 1%, or 3% formulation of OPA-15406 ointment as a single dose. We assess the AUC12h x of OPA-15406.
Time Frame: Baseline, 2 ,3, 4, 8, 10, 12, 16, 24 and 48 hrs
Measure: Mean (Standard Deviation); unit: ng･h/mL
Arm/Group | 0.3% OPA-15406 Ointment in a Single Administration Period | 1% OPA-15406 Ointment in a Single Administration Period | 3% OPA-15406 Ointment in a Single Administration Period
Number analyzed (Participants) | 8 | 8 | 8
ng･h/mL | 3.74 (2.32) | 6.42 (4.86) | 11.2 (6.24)

4. Secondary Outcome: AUC12h of OPA-15406 in the Multiple Administration Period
Description: as for outcome 2
Time Frame: Baseline, 2 ,3, 4, 8, 10, 12, 16, 24 and 48 hrs at Day 14
Measure: Mean (Standard Deviation); unit: ng･h/mL
Arm/Group | 0.3 % OPA-15406 Ointment in the Multiple Administration Period | 1 % OPA-15406 Ointment in the Multiple Administration Period | 3% OPA-15406 Ointment in the Multiple Administration Period
Number analyzed (Participants) | 8 | 8 | 8
ng･h/mL | 4.65 (3.07) | 7.84 (1.78) | 16.6 (4.99)

ADVERSE EVENTS:
Time Frame: A single administration: From date of informed consent to 48 hours post dose The multiple administration: From date of assigned IMP twice daily to 16 days post dose
Groups:
- 0.3 % OPA-15406 Ointment in a Single Administration Period: 32 subjects were randomly allocated to 4 treatment groups (8 subjects per dose). In a single administration period, same subjects were treated with assigned 0.3% OPA-15406 ointment
- 1% OPA-15406 Ointment in a Single Administaration Period: 32 subjects were randomly allocated to 4 treatment groups (8 subjects per dose). In a single and administration period, same subjects were treated with assigned 1% OPA-15406 ointment.
- 3% OPA-15406 Ointment in a Single Administaration Period: 32 subjects were randomly allocated to 4 treatment groups (8 subjects per dose). In a single administration period, same subjects were treated with assigned 3% OPA-15406 ointment.
- Placebo in a Single Adminstaration Period: 32 subjects were randomly allocated to 4 treatment groups (8 subjects per dose). In a single administration period, same subjects were treated with assigned placebo ointment.
- 0.3 % OPA-15406 Ointment in the Multiple Administration Period: In the multiple administration period, same subjects were treated with assigned 0.3 % OPA-15406 ointment twice daily for 14 days and assessed until 48 hours post dose.
- 1 % OPA-15406 Ointment in the Multiple Administration Period: In the multiple administration period, same subjects were treated with assigned 1 % OPA-15406 ointment twice daily for 14 days and assessed until 48 hours post dose.
- 3 % OPA-15406 Ointment in the Multiple Administration Period: In the multiple administration period, same subjects were treated with assigned 3 % OPA-15406 ointment twice daily for 14 days and assessed until 48 hours post dose.
- Placebo Ointment in the Multiple Administration Period: In the multiple administration period, same subjects were treated with assigned placebo ointment twice daily for 14 days and assessed until 48 hours post dose.
Arm/Group | 0.3 % OPA-15406 Ointment in a Single Administration Period | 1% OPA-15406 Ointment in a Single Administaration Period | 3% OPA-15406 Ointment in a Single Administaration Period | Placebo in a Single Adminstaration Period | 0.3 % OPA-15406 Ointment in the Multiple Administration Period | 1 % OPA-15406 Ointment in the Multiple Administration Period | 3 % OPA-15406 Ointment in the Multiple Administration Period | Placebo Ointment in the Multiple Administration Period
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No